CLINICAL TRIAL: NCT02579798
Title: Does Pulmonary Compliance Optimization Through PEEP Manipulations Reduces the Incidence of Postoperative Hypoxaemia in Bariatric Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Philippe VAN DER LINDEN, Head of clinic, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHUB-CRF
Record Dates: First submitted 2015-10-12; First posted 2015-10-20 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Bariatric Surgery
Keywords: Bariatric surgery; Post-surgery hypoxemia; Obesity
MeSH Terms: conditions — Obesity | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEP 10 cmH20 (Experimental): In this group, a PEEP of 10 cmH20 is applied for the duration of the intervention and a recruitment maneuver is applied each time the SpO2 (oxygen pulsated saturation) drops below 95%.
  Interventions: Device: PEEP (positive end-expiratory pressure)
- optimal PEEP (Active Comparator): In this group, 10 cmH20 PEEP is applied immediately. Then the "optimal PEEP" is sought at three key moments. It is determined by the best value of lung compliance found in the patient. It is sought by increasing or decreasing the value of the PEEP by increments or decrements of 2 cmH20. If after 6 respiratory cycles, the value of the compliance is increased, the investigator continues to increase the value of the PEEP. On the other hand, if the value of compliance is reduced, the investigator reduces the value of PEEP. The value of the PEEP selected shall in no event exceed the set pressure range (maximum pressure plate of 30 cmH20 and maximum inspiratory peak pressure 40cmH20). A recruitment maneuver is applied each time the SpO2 drops below 95%, as in the PEEP 10cmH2O group.
  Interventions: Device: PEEP (positive end-expiratory pressure)

INTERVENTIONS:
Device: PEEP (positive end-expiratory pressure)

SUMMARY:
General anesthesia, even in patients in good health, impairs gas exchanges and ventilatory mechanics. These effects result primarily from atelectasis formation. They occur in 85-90% of healthy patients in the minutes following the induction when a positive end expiratory pressure (PEEP) is not used.

The functional residual capacity (FRC) of obese patients during general anesthesia is even smaller than the one of healthy patients. There is a direct relationship between the body mass index and the decrease of the functional residual capacity. Obese patients have therefore more atelectasis. The increased abdominal pressure during the pneumoperitoneum will increase the decrease of the CRF, and thus aggravate the formation of these atelectasis.

Atelectasis affect the peroperative gas exchanges and are likely to be involved in the worsening of postoperative hypoxemia episodes. In addition, atelectasis alter the clearance of secretions and the lymph flow, which predispose to lung infections.Taking all these factors into account, it is logical to think that the atelectasis presence can lead to an increase of the postsurgical morbidity (respiratory distress, infections). That is why actively fighting against the formation of these atelectasis is important.

There is a lack of scientific evidence to say that the strategies against atelectasis as PEEP have a significant impact on the patient's postoperative status. The expected clinical benefits balance (reduction of respiratory distress episodes, infections and mortality) versus the risks linked to the maneuvers done to reduce the development of atelectasis (barotraumas, cardiac complications) remains to be determined.

The primary goal of this study is to evaluate the impact of two different alveolar recruitment strategies on the incidence of postoperative hypoxemia in obese patients after bariatric surgery.

The secondary objectives of this study are to compare the number of recruitment maneuvers, the Pa02 / FI02 ratio (ratio of arterial oxygen partial pressure to fractional inspired oxygen), the dynamic compliance, the anatomic dead space and intraoperative PaCO2-EtCO2 gradient (arterial and end tidal gradient) between two alveolar recruitment strategies applied in obese patients during laparoscopic bariatric surgery (gastric bypass or sleeve gastrectomy).

The tertiary objectives of this study are to report the number of respiratory complications and postoperative wound infections at the 30th postoperative day.

DETAILED DESCRIPTION:
General anesthesia, even in patients in good health, impairs gas exchanges and ventilatory mechanics. These effects result primarily from atelectasis formation. They occur in 85-90% of healthy patients in the minutes following the induction when a positive end expiratory pressure (PEEP) is not used.

These atelectasis are formed on one hand by the reduction of the functional residual capacity (FRC) following a compression mechanism (loss of the inspiratory muscle tone, which is accompanied by a chest wall configuration change and a diaphragm cephalic movement) and on the other hand by a denitrogenation absorption process (ventilation at high Fi02 (oxygen inspired fraction) causing complete absorption of O2 with lack of support for the alveolus, which then collapses).

The FRC of obese patients during general anesthesia is even smaller than the one of healthy patients. There is a direct relationship between the body mass index and the decrease of the functional residual capacity. Obese patients have therefore more atelectasis. The increased abdominal pressure during the pneumoperitoneum will increase the decrease of the CRF, and thus aggravate the formation of these atelectasis.

Atelectasis affect the peroperative gas exchanges and are likely to be involved in the worsening of postoperative hypoxemia episodes. In addition, atelectasis alter the clearance of secretions and the lymph flow, which predispose to lung infections.Taking all these factors into account, it is logical to think that the atelectasis presence can lead to an increase of the postsurgical morbidity (respiratory distress, infections). That is why actively fighting against the formation of these atelectasis is important.

Several strategies have been studied in order to improve respiratory mechanics and reduce impaired gas exchange during laparoscopic surgery in obese patients. The position called "chair", mechanical ventilation with PEEP, recruitment maneuvers followed by the PEEP, and spontaneous ventilation with CPAP before extubation, are all strategies that have proven effective to decrease development these atelectasis.

Currently, the scientific community agrees on the fact that PEEP improves intraoperative respiratory function (improved compliance, oxygenation) especially in conjunction with recruitment maneuvers.

But there is a lack of scientific evidence to say that the strategies against atelectasis as PEEP have a significant impact on the patient's postoperative status. The expected clinical benefits balance (reduction of respiratory distress episodes, infections and mortality) versus the risks linked to the maneuvers done to reduce the development of atelectasis (barotraumas, cardiac complications) remains to be determined.

The primary goal of this study is to evaluate the impact of two different alveolar recruitment strategies on the incidence of postoperative hypoxemia in obese patients after bariatric surgery.

The secondary objectives of this study are to compare the number of recruitment maneuvers, the Pa02 / FI02 ratio, the dynamic compliance, the anatomic dead space and intraoperative PaCO2-EtCO2 gradient between two alveolar recruitment strategies applied in obese patients during laparoscopic bariatric surgery (gastric bypass or sleeve gastrectomy).

The tertiary objectives of this study are to report the number of respiratory complications and postoperative wound infections at the 30th postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* ASA score (American Society of Anesthesiologists ) of II or III
* BMI > 35 kg/m²
* Elective laparoscopic bariatric surgery: gastric bypass or sleeve

Exclusion Criteria:

* Restrictive (CPT <65%) or obstructive (VEMS/CV < 69%) chronic lung disease
* Increase of the intracranial pressure
* History of smoking with chronic obstructive disease (VEMS/CV)
* Active tabagism
* Ongoing pregnancy
* History of heart failure (NYHA III or IV) or coronary artery disease
* Urgent surgery
* Allergy to a drug used within the study
* Lack of written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of hypoxemia episodes (Sp02<90%) | continuously during 48h after surgery
  This will be monitored by a portable saturometer (OxyTrue A, Bluepoint, Germany). This saturometer will allow the investigators to count the number of hypoxemia episodes (Sp02<90%) and their duration in obese patients, in the postoperative period.
Number of hypoxemia episodes (Sp02<95%) | continuously during 48h after surgery
  This will be monitored by a portable saturometer (OxyTrue A, Bluepoint, Germany). This saturometer will allow the investigators to count the number of hypoxemia episodes (Sp02<95%) and their duration in obese patients, in the postoperative period.

SECONDARY OUTCOMES:
Number of recruitment manoeuvers | From the beginning of the surgery till moment 1 (after induction/intubation, patient laying flat, without pneumoperitoneum)
  Recruitment manoeuver are performed if patient saturation drops below 95%.
Number of recruitment manoeuvers | From moment 1 till moment 2 (after peritoneal insufflation and anti-trendenlenbourg (anti-trent) implementation)
  Recruitment manoeuver are performed if patient saturation drops below 95%.
Number of recruitment manoeuvers | From moment 2 till moment 3 (after pneumoperitoneum exsufflation - patient lying flat)
  Recruitment manoeuver are performed if patient saturation drops below 95%.
Number of recruitment manoeuvers | From moment 3 till the end of the surgery (patient leaving the theater)
  Recruitment manoeuver are performed if patient saturation drops below 95%.
Pulmonary dynamic compliance (Cd) - preoperative | Just before surgery, at ambient air contact
  This will be determined by the following formula: Cd = Vt/P(peak)-PEEP and expressed in mL/cmH2O
Pulmonary dynamic compliance (Cd) - moment 1 | just after the anesthesia induction/intubation, patient laying flat, without pneumoperitory
  This will be determined by the following formula: Cd = Vt/P(peak)-PEEP and expressed in mL/cmH2O
Pulmonary dynamic compliance (Cd) -moment 2 | just after peritoneal insufflation and anti-trendenlenbourg (anti-trent) implementation
  This will be determined by the following formula: Cd = Vt/P(peak)-PEEP and expressed in mL/cmH2O
Pulmonary dynamic compliance (Cd) -moment 3 | just after pneumoperitoneum exsufflation - patient lying flat
  This will be determined by the following formula: Cd = Vt/P(peak)-PEEP and expressed in mL/cmH2O
Pulmonary dynamic compliance (Cd) -if recruitment manoeuvers | Five minutes after any recruitment manoeuver
  This will be determined by the following formula: Cd = Vt/P(peak)-PEEP and expressed in mL/cmH2O
Anatomic dead space - preoperative | Just before surgery, at ambient air contact
  This will be determined by this formula: VD = VT (1-PEtCO2/PaC02)
Anatomic dead space -moment 1 | just after the anesthesia induction/intubation, patient laying flat, without pneumoperitory
  This will be determined by this formula: VD = VT (1-PEtCO2/PaC02)
Anatomic dead space -moment 2 | just after peritoneal insufflation and anti-trendenlenbourg (anti-trent) implementation
  This will be determined by this formula: VD = VT (1-PEtCO2/PaC02)
Anatomic dead space -moment 3 | just after pneumoperitoneum exsufflation - patient lying flat
  This will be determined by this formula: VD = VT (1-PEtCO2/PaC02)
Anatomic dead space -if recruitment manoeuvers | Five minutes after any recruitment manoeuver
  This will be determined by this formula: VD = VT (1-PEtCO2/PaC02)
PaO2/FiO2 ratio - preoperative | Just before surgery, at ambient air contact
  Arterial oxygen partial pressure to fractional inspired oxygen ratio
PaO2/FiO2 ratio - moment 1 | just after the anesthesia induction/intubation, patient laying flat, without pneumoperitory
  Arterial oxygen partial pressure to fractional inspired oxygen ratio
PaO2/FiO2 ratio - moment 2 | just after peritoneal insufflation and anti-trendenlenbourg (anti-trent) implementation
  Arterial oxygen partial pressure to fractional inspired oxygen ratio
PaO2/FiO2 ratio - moment 3 | just after pneumoperitoneum exsufflation - patient lying flat
  Arterial oxygen partial pressure to fractional inspired oxygen ratio
PaO2/FiO2 ratio - if recruitment manoeuvers | Five minutes after any recruitment manoeuver
  Arterial oxygen partial pressure to fractional inspired oxygen ratio
PaCO2-EtCO2 gradient - preoperative | Just before surgery, at ambient air contact
  The gradient between the partial pressure of carbon dioxide in the arterial blood (PaCO2) and the CO2 end-tidal partial pressure (EtCO2) is used to evaluate the effectiveness of alveolar recruitment.
PaCO2-EtCO2 gradient - moment 1 | just after the anesthesia induction/intubation, patient laying flat, without pneumoperitory
  The gradient between the partial pressure of carbon dioxide in the arterial blood (PaCO2) and the CO2 end-tidal partial pressure (EtCO2) is used to evaluate the effectiveness of alveolar recruitment.
PaCO2-EtCO2 gradient - moment 2 | just after peritoneal insufflation and anti-trendenlenbourg (anti-trent) implementation
  The gradient between the partial pressure of carbon dioxide in the arterial blood (PaCO2) and the CO2 end-tidal partial pressure (EtCO2) is used to evaluate the effectiveness of alveolar recruitment.
PaCO2-EtCO2 gradient - moment 3 | just after pneumoperitoneum exsufflation - patient lying flat
  The gradient between the partial pressure of carbon dioxide in the arterial blood (PaCO2) and the CO2 end-tidal partial pressure (EtCO2) is used to evaluate the effectiveness of alveolar recruitment.
PaCO2-EtCO2 gradient - if recruitment manoeuvers | Five minutes after any recruitment manoeuver
  The gradient between the partial pressure of carbon dioxide in the arterial blood (PaCO2) and the CO2 end-tidal partial pressure (EtCO2) is used to evaluate the effectiveness of alveolar recruitment.
Number of respiratory complications | 30 days after surgery
  Number of hospitalisations due to respiratory complications within 30 days after surgery.
Number of postoperative wound infections | 30 days after surgery
  All patients are seen at the surgical consultation on day 30 after surgery. The anamnesis performed during that consultation enables the investigators to identify patients with wound infections (defined as a need for local or oral antibiotics, additional hospitalisation or abnormal cicatrisation).
Pre-operative physiologic measures: cardiac frequency (FC) | Just before surgery, at ambient air contact
  The hemodynamic and respiratory parameters of the patient are measured by means of a Datex-Ohmeda Acertys machine (Aisys type).
Pre-operative physiologic measures: Arterial tension (TA) | Just before surgery, at ambient air contact
  The hemodynamic and respiratory parameters of the patient are measured by means of a Datex-Ohmeda Acertys machine (Aisys type).
Pre-operative physiologic measures: pH | Just before surgery, at ambient air contact
  The hemodynamic and respiratory parameters of the patient are measured by means of a Datex-Ohmeda Acertys machine (Aisys type).
Pre-operative physiologic measures: partial pressure of carbon dioxide in the arterial blood (PaCO2) | Just before surgery, at ambient air contact
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens).
Operative physiologic measures - moment 1: FC | just after induction/intubation, patient laying flat, without pneumoperitoneum
  The hemodynamic and respiratory parameters of the patient are measured by means of a Datex-Ohmeda Acertys machine (Aisys type).
Operative physiologic measures - moment 1: PAM (Average arterial pressure) | just after induction/intubation, patient laying flat, without pneumoperitoneum
  The hemodynamic and respiratory parameters of the patient are measured by means of a Datex-Ohmeda Acertys machine (Aisys type).
Operative physiologic measures - moment 1: pH | just after induction/intubation, patient laying flat, without pneumoperitoneum
  The hemodynamic and respiratory parameters of the patient are measured by means of a Datex-Ohmeda Acertys machine (Aisys type).
Operative physiologic measures - moment 1: PaCO2 | just after induction/intubation, patient laying flat, without pneumoperitoneum
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Operative physiologic measures - moment 1: CO2 | just after induction/intubation, patient laying flat, without pneumoperitoneum
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Operative physiologic measures - moment 2: FC | just after peritoneal insufflation and anti-trendenlenbourg (anti-trent) implementation
  The hemodynamic and respiratory parameters of the patient are measured by means of a Datex-Ohmeda Acertys machine (Aisys type).
Operative physiologic measures - moment 2: PAM | just after peritoneal insufflation and anti-trendenlenbourg (anti-trent) implementation
  The hemodynamic and respiratory parameters of the patient are measured by means of a Datex-Ohmeda Acertys machine (Aisys type).
Operative physiologic measures - moment 2: pH | just after peritoneal insufflation and anti-trendenlenbourg (anti-trent) implementation
  The hemodynamic and respiratory parameters of the patient are measured by means of a Datex-Ohmeda Acertys machine (Aisys type).
Operative physiologic measures - moment 2: PaCO2 | just after peritoneal insufflation and anti-trendenlenbourg (anti-trent) implementation
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Operative physiologic measures - moment 2: CO2 | just after peritoneal insufflation and anti-trendenlenbourg (anti-trent) implementation
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Operative physiologic measures - moment 3: FC | just after pneumoperitoneum exsufflation - patient lying flat
  The hemodynamic and respiratory parameters of the patient are measured by means of a Datex-Ohmeda Acertys machine (Aisys type).
Operative physiologic measures - moment 3: PAM | just after pneumoperitoneum exsufflation - patient lying flat
  The hemodynamic and respiratory parameters of the patient are measured by means of a Datex-Ohmeda Acertys machine (Aisys type).
Operative physiologic measures - moment 3: pH | just after pneumoperitoneum exsufflation - patient lying flat
  The hemodynamic and respiratory parameters of the patient are measured by means of a Datex-Ohmeda Acertys machine (Aisys type).
Operative physiologic measures - moment 3: CO2 | just after pneumoperitoneum exsufflation - patient lying flat
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Operative physiologic measures - moment 3: PaCO2 | just after pneumoperitoneum exsufflation - patient lying flat
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Operative physiologic measures - if recruitment manoeuvers occurs: FC | Five minutes after any recruitment manoeuver
  The hemodynamic and respiratory parameters of the patient are measured by means of a Datex-Ohmeda Acertys machine (Aisys type).
Operative physiologic measures - if recruitment manoeuvers occurs: PAM | Five minutes after any recruitment manoeuver
  The hemodynamic and respiratory parameters of the patient are measured by means of a Datex-Ohmeda Acertys machine (Aisys type).
Operative physiologic measures - if recruitment manoeuvers occurs: SpO2 | Five minutes after any recruitment manoeuver
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Operative physiologic measures - if recruitment manoeuvers occurs: pH | Five minutes after any recruitment manoeuver
  The hemodynamic and respiratory parameters of the patient are measured by means of a Datex-Ohmeda Acertys machine (Aisys type).
Operative physiologic measures - if recruitment manoeuvers occurs: PaCO2 | Five minutes after any recruitment manoeuver
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Operative physiologic measures - if recruitment manoeuvers occurs: PaO2 | Five minutes after any recruitment manoeuver
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Operative physiologic measures - if recruitment manoeuvers occurs: CO2 | Five minutes after any recruitment manoeuver
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Pre-operative physiologic measures: partial pressure of oxygen in the arterial blood (PaO2) | Just before surgery, at ambient air contact
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Operative physiologic measures - moment 1: PaO2 | just after induction/intubation, patient laying flat, without pneumoperitoneum
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Operative physiologic measures - moment 2: PaO2 | just after peritoneal insufflation and anti-trendenlenbourg (anti-trent) implementation
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Operative physiologic measures - moment 3: PaO2 | just after pneumoperitoneum exsufflation - patient lying flat
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Pre-operative physiologic measures: Oxygen Pulsated Saturation (SpO2) | Just before surgery, at ambient air contact
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Operative physiologic measures - moment 1: SpO2 | just after induction/intubation, patient laying flat, without pneumoperitoneum
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Operative physiologic measures - moment 2: SpO2 | just after peritoneal insufflation and anti-trendenlenbourg (anti-trent) implementation
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)
Operative physiologic measures - moment 3: SpO2 | just after pneumoperitoneum exsufflation - patient lying flat
  The gasometric parameters of the patient are analyzed with a Rapidlab 1265 machine (Siemens)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Van der Linden, MD, Principal Investigator — CHU Brugmann; Van Hecke Delphine, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Coussa M, Proietti S, Schnyder P, Frascarolo P, Suter M, Spahn DR, Magnusson L. Prevention of atelectasis formation during the induction of general anesthesia in morbidly obese patients. Anesth Analg. 2004 May;98(5):1491-5, table of contents. doi: 10.1213/01.ane.0000111743.61132.99. PMID 15105237
- [Background] Imberger G, McIlroy D, Pace NL, Wetterslev J, Brok J, Moller AM. Positive end-expiratory pressure (PEEP) during anaesthesia for the prevention of mortality and postoperative pulmonary complications. Cochrane Database Syst Rev. 2010 Sep 8;(9):CD007922. doi: 10.1002/14651858.CD007922.pub2. PMID 20824871
- [Background] Eichenberger A, Proietti S, Wicky S, Frascarolo P, Suter M, Spahn DR, Magnusson L. Morbid obesity and postoperative pulmonary atelectasis: an underestimated problem. Anesth Analg. 2002 Dec;95(6):1788-92, table of contents. doi: 10.1097/00000539-200212000-00060. PMID 12456460
- [Background] Whalen FX, Gajic O, Thompson GB, Kendrick ML, Que FL, Williams BA, Joyner MJ, Hubmayr RD, Warner DO, Sprung J. The effects of the alveolar recruitment maneuver and positive end-expiratory pressure on arterial oxygenation during laparoscopic bariatric surgery. Anesth Analg. 2006 Jan;102(1):298-305. doi: 10.1213/01.ane.0000183655.57275.7a. PMID 16368847
- [Background] Futier E, Constantin JM, Pelosi P, Chanques G, Kwiatkoskwi F, Jaber S, Bazin JE. Intraoperative recruitment maneuver reverses detrimental pneumoperitoneum-induced respiratory effects in healthy weight and obese patients undergoing laparoscopy. Anesthesiology. 2010 Dec;113(6):1310-9. doi: 10.1097/ALN.0b013e3181fc640a. PMID 21068660
- [Background] Almarakbi WA, Fawzi HM, Alhashemi JA. Effects of four intraoperative ventilatory strategies on respiratory compliance and gas exchange during laparoscopic gastric banding in obese patients. Br J Anaesth. 2009 Jun;102(6):862-8. doi: 10.1093/bja/aep084. Epub 2009 Apr 29. PMID 19403595
- [Background] Reinius H, Jonsson L, Gustafsson S, Sundbom M, Duvernoy O, Pelosi P, Hedenstierna G, Freden F. Prevention of atelectasis in morbidly obese patients during general anesthesia and paralysis: a computerized tomography study. Anesthesiology. 2009 Nov;111(5):979-87. doi: 10.1097/ALN.0b013e3181b87edb. PMID 19809292
- [Background] Pelosi P, Ravagnan I, Giurati G, Panigada M, Bottino N, Tredici S, Eccher G, Gattinoni L. Positive end-expiratory pressure improves respiratory function in obese but not in normal subjects during anesthesia and paralysis. Anesthesiology. 1999 Nov;91(5):1221-31. doi: 10.1097/00000542-199911000-00011. PMID 10551570
- [Background] Tusman G, Bohm SH, Suarez-Sipmann F, Turchetto E. Alveolar recruitment improves ventilatory efficiency of the lungs during anesthesia. Can J Anaesth. 2004 Aug-Sep;51(7):723-7. doi: 10.1007/BF03018433. PMID 15310643
- [Background] Maisch S, Reissmann H, Fuellekrug B, Weismann D, Rutkowski T, Tusman G, Bohm SH. Compliance and dead space fraction indicate an optimal level of positive end-expiratory pressure after recruitment in anesthetized patients. Anesth Analg. 2008 Jan;106(1):175-81, table of contents. doi: 10.1213/01.ane.0000287684.74505.49. PMID 18165575
- [Background] Strang CM, Hachenberg T, Freden F, Hedenstierna G. Development of atelectasis and arterial to end-tidal PCO2-difference in a porcine model of pneumoperitoneum. Br J Anaesth. 2009 Aug;103(2):298-303. doi: 10.1093/bja/aep102. Epub 2009 May 13. PMID 19443420
- [Background] Gander S, Frascarolo P, Suter M, Spahn DR, Magnusson L. Positive end-expiratory pressure during induction of general anesthesia increases duration of nonhypoxic apnea in morbidly obese patients. Anesth Analg. 2005 Feb;100(2):580-584. doi: 10.1213/01.ANE.0000143339.40385.1B. PMID 15673897
- [Background] Hans GA, Sottiaux TM, Lamy ML, Joris JL. Ventilatory management during routine general anaesthesia. Eur J Anaesthesiol. 2009 Jan;26(1):1-8. doi: 10.1097/EJA.0b000e000000f1fb. PMID 19122544
- [Background] Mercat A, Richard JC, Vielle B, Jaber S, Osman D, Diehl JL, Lefrant JY, Prat G, Richecoeur J, Nieszkowska A, Gervais C, Baudot J, Bouadma L, Brochard L; Expiratory Pressure (Express) Study Group. Positive end-expiratory pressure setting in adults with acute lung injury and acute respiratory distress syndrome: a randomized controlled trial. JAMA. 2008 Feb 13;299(6):646-55. doi: 10.1001/jama.299.6.646. PMID 18270353
- [Background] Gattinoni L, Carlesso E, Brazzi L, Caironi P. Positive end-expiratory pressure. Curr Opin Crit Care. 2010 Feb;16(1):39-44. doi: 10.1097/MCC.0b013e3283354723. PMID 19996966
- [Derived] Van Hecke D, Bidgoli JS, Van der Linden P. Does Lung Compliance Optimization Through PEEP Manipulations Reduce the Incidence of Postoperative Hypoxemia in Laparoscopic Bariatric Surgery? A Randomized Trial. Obes Surg. 2019 Apr;29(4):1268-1275. doi: 10.1007/s11695-018-03662-x. PMID 30612327